CLINICAL TRIAL: NCT00005614
Title: Management of Metastatic Breast Cancer in Frail Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11909; NCI-G00-1748 (Other: NCI)
Record Dates: First submitted 2000-05-02; First posted 2004-07-26 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine Treatment (Experimental): Patients receive gemcitabine IV over 1 hour weekly for 7 consecutive weeks in an 8 week course. Treatment then continues weekly for 3 consecutive weeks in 4 week courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed prior to treatment and then every 12 weeks. Patients are followed every 3 months for 2 years, then every 6 months until year 5, and then annually thereafter.
  Interventions: Drug: Gemcitabine hydrochloride

INTERVENTIONS:
Drug: Gemcitabine hydrochloride — Gemcitabine via IV
  Other Names: Gemzar

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine in treating elderly women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and efficacy of gemcitabine in the treatment of elderly women with metastatic breast cancer. II. Evaluate the quality of life in these patients.

OUTLINE: Patients receive gemcitabine IV over 1 hour weekly for 7 consecutive weeks in an 8 week course. Treatment then continues weekly for 3 consecutive weeks in 4 week courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed prior to treatment and then every 12 weeks. Patients are followed every 3 months for 2 years, then every 6 months until year 5, and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Metastatic breast cancer Measurable disease No progression after 3 or more different forms of chemotherapy Hormone receptor positive breast cancer must be refractory to at least two forms of hormonal treatment (including antiestrogen, aromatase inhibitor, and/or progestin) unless there is life threatening metastases (e.g., lymphangitic metastases to the lung or liver metastases) Must meet at least one of the following characteristics for frailty: ECOG 2-4 Dependence in at least one activity of daily living 85 and over History of three or more falls in the past 6 months Mild dementia (must be oriented in time, space, and location) Three or more comorbid conditions Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 65 and over Sex: Female Menopausal status: Not specified Performance status: See Disease Characteristics Life expectancy: Greater than 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Neutropenia or thrombocytopenia secondary to myelophthisis from breast cancer allowed Hepatic: Increased bilirubin allowed Renal: Renal insufficiency allowed Cardiovascular: Congestive heart failure allowed Other: No known allergy to gemcitabine

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: See Disease Characteristics Radiotherapy: At least 4 weeks since prior radiotherapy to bony areas or CNS metastases Surgery: Not specified Other: Concurrent bisphosphonates allowed No concurrent participation in other investigational studies

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-08; Primary Completion 2000-06 (Actual); Study Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Investigators planned to determine efficacy (objective response rate [ORR] by Response Evaluation Criteria In Solid Tumors [RECIST]).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 2 years
  Investigators planned to review adverse events utilizing Common Toxicity Criteria (CTC) V3.

CONTACTS AND LOCATIONS:
Overall Officials: Lodovico Balducci, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute